CLINICAL TRIAL: NCT02634463
Title: Whole Blood and Plasma Sample Collection for the Development of Antipsychotic Immunoassays From Participants Taking Aripiprazole, Olanzapine, Paliperidone, or Risperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108047; CODX0001-NAP-1004 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2015-11-02; First posted 2015-12-18 (Estimated); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Immunoassay; Antipsychotic
Keywords: Immunoassay; Antipsychotic; Aripiprazole; Olanzapine; Paliperidone; Risperidone
MeSH Terms: interventions — Aripiprazole; Olanzapine; Paliperidone Palmitate; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Antipsychotic Immunoassay Development Participants (Other): No study agent will be administered as a part of this study. Participants must be on Aripiprazole or Olanzapine, or Paliperidone or Risperidone, orally, daily or long-acting injectable versions, as part of the treatment for a psychiatric illness to be eligible for enrollment in this study. Whole Blood and Plasma Samples will be collected for use in the development of antipsychotic immunoassays. Participants may also be on long acting injectable versions of the medication.
  Interventions: Drug: Aripiprazole; Other: Olanzapine; Drug: Paliperidone; Drug: Risperidone

INTERVENTIONS:
Drug: Aripiprazole — No study agent will be administered as a part of this study. Participants must be on Aripiprazole 5 milligram (mg) (minimum dose) to 30 mg (maximum dose), orally, daily or long-acting injectable versions (300-400 mg once every 4 weeks), as part of the treatment for a psychiatric illness to be eligible for enrollment in this study. Whole Blood and Plasma Samples will be collected for development of antipsychotic immunoassays.
Other: Olanzapine — No study agent will be administered as a part of this study. Participants must be on Olanzapine 5 mg (minimum dose) to 30 mg (maximum dose), orally, daily or long-acting injectable versions (150-405 mg once every 2-4 weeks), as part of the treatment for a psychiatric illness to be eligible for enrollment in this study. Whole Blood and Plasma Samples will be collected for Development of the antipsychotic immunoassays.
Drug: Paliperidone — No study agent will be administered as a part of this study. Participants must be on Paliperidone 3 mg (minimum dose) to 12 mg (maximum dose), orally, daily or long-acting injectable versions (25-150 mg equivalent [eq.] once every 4 weeks), as part of the treatment for a psychiatric illness to be eligible for enrollment in this study. Whole Blood and Plasma Samples will be collected for Development of the antipsychotic immunoassays.
Drug: Risperidone — No study agent will be administered as a part of this study. Participants must be on Risperidone 1 mg (minimum dose) to 8 mg (maximum dose), orally, daily or long-acting injectable versions (12.5-50 mg once every 2 weeks), as part of the treatment for a psychiatric illness to be eligible for enrollment in this study. Whole Blood and Plasma Samples will be collected for Development of the antipsychotic immunoassays.

SUMMARY:
The purpose of this study is to collect whole blood and plasma venous and capillary samples from participants taking aripiprazole, olanzapine, paliperidone, or risperidone for the development of antipsychotic immunoassays.

DETAILED DESCRIPTION:
This is a Phase 0, multicenter (when more than one hospital work on a medical research study) study including participants taking aripiprazole, olanzapine, paliperidone or risperidone. Participants will provide blood samples to be used in development of antipsychotic immunoassays. At different times, assay development will require venous, capillary, or both types of blood samples. Overall, at a single study visit, a minimum of approximately 0.1 milliliter (mL) to a maximum of approximately 15 mL of blood will be collected from all sources. Across all study visits, a maximum of 450 mL of blood will be collected from a participant. The frequency of collections (study visits) will depend on the needs of assay development. A particular participant may participate for only 1 sample collection or multiple sample collections (study visits). This study will continue for an indefinite period of time. The participant's direct involvement in the study will be continued until the study is ended, the participant has given 450 mL of blood, or the participant withdraws consent or is excluded from participation for medical and/or inclusion/exclusion criteria reasons. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 18 years of age
* Must be taking one or more of the following antipsychotic medications: aripiprazole, olanzapine, paliperidone, and/or risperidone as part of the treatment for a psychiatric illness
* Must be psychiatrically stable as determined by their psychiatrist or similar clinician. The participant must not have had suicidal behavior or clinically significant suicidal ideation during the week prior to Screening, according to the investigator's judgment
* Generally healthy and has no clinically significant or unstable medical problems as determined by the investigator, except for the indication for which the antipsychotic treatment is being prescribed. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study. Consent cannot be given by a guardian or other person

Exclusion Criteria:

* Participants who regularly miss more than one dose of antipsychotic medication in a typical week
* During Screening or during the conduct of the study, the participant has an active substance use disorder of moderate or severe intensity except for tobacco (Diagnostic and Statistical Manual of Mental Disorders [DSM-5] definition) or acute intoxication at any study visit as determined by the investigator
* Donated blood or had blood loss of greater than (>) 450 milliliter (mL) in the past 3 months. Participants may not donate blood during participation in the study
* Any participant who has had a surgical and/ or biopsy procedure within the last 6 weeks. For enrolled participants, additional study-related blood draws will need to be delayed for at least 6 weeks after such a procedure or significant blood loss
* Any participant who has had a negative reaction to a blood draw (such as fainting) in the past

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2016-11-09 (Actual); Study Completion 2016-11-09 (Actual)

PRIMARY OUTCOMES:
Immunoassay Antipsychotic In Blood | Up to 1 year
  Whole blood and plasma venous and capillary samples will be collected from participants taking aripiprazole, olanzapine, paliperidone, or risperidone to determine the concentration, which will be used in the development of antipsychotic immunoassays.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Duffel, Belgium